CLINICAL TRIAL: NCT04566146
Title: A Clinical Prediction Rule to Identify Patients With Shoulder Impingement Syndrome Response to Scapular Training
Brief Title: Clinical Prediction Rule for Patients With Shoulder Impingement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hager Tarek Khater Mohamed, demonestrator in the department of physical therapy for musculoskeletal disorders and its surgery, faculty of physical therapy, cairo university, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CPR for patients with SIS
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Physical Therapy
Keywords: clinical prediction rule; shoulder impingement syndrome; subacromial impingement syndrome; scapular training
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 45 patients with subacromial impingement syndrome (Other): Forty-five patients between the age 18 and 45 years old, will be referred by orthopaedist as subacromial impingement syndrome (stage Ⅰ and ⅠⅠ Neer's classification)
  Interventions: Other: scapular muscle training, serratus anterior strength, scapular stabilization exercises

INTERVENTIONS:
Other: scapular muscle training, serratus anterior strength, scapular stabilization exercises — patients will be scheduled to attend physical therapy three sessions per week for one month. Three sets of 10 repetitions for each exercise were prescribed per session, with a 1-minute rest between sets.

SUMMARY:
To investigate if pain severity, scapular upward rotation angle and upper trapezius/serratus anterior isometric strength ratio can predict patient's response to scapular training in patients with subacromial impingement syndrome.

DETAILED DESCRIPTION:
Shoulder impingement syndrome (SIS) is the most commonly diagnosed shoulder disorder. In literature shoulder impingement is reported between 48% and 65% of all painful shoulder conditions.

The coordinated coupled motion between the scapula and humerus, the so-called scapulohumeral rhythm (SHR), is needed for efficient arm movement. Reduced scapular mobility reduces the acromio-humeral distance during arm abduction and therefore increases the risk for shoulder impingement syndrome.

Clinical prediction rules (CPRs) are tools designed to improve decision making in clinical practice by assisting practitioners in making a particular diagnosis, establishing a prognosis, or matching patients to optimal interventions based on a parsimonious subset of predictor variables from the history and physical examination.

HYPOTHESES:

Pain severity will not be predictor for treatment success in patients suffering from subacromial impingement syndrome treated with scapular training.

Scapular upward rotation angle will not be predictor for treatment success in patients suffering from subacromial impingement syndrome treated with scapular training.

Ratio of upper trapezius /serratus anterior isometric strength will not be predictor for treatment success in patients suffering from subacromial impingement syndrome treated with scapular training.

RESEARCH QUESTION:

Does pain severity, scapular upward rotation angle and upper trapezius/serratus anterior isometric strength ratio predict patient's esponse to scapular training in patients with subacromial impingement syndrome?

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-45 years old patients diagnosed as subacromial impingement syndrome.
* 2. Patients will be included in this study if they have at least 3 of the following 6 criteria:
* 2a. Positive "Neer sign": The examiner passively flexes the humerus with medial rotation to end-range with over pressure. The patient's facial expression and the reproduction of the pain confirm the presence of impingement.
* 2b. Positive "Hawkins sign": The shoulder is passively placed in approximately 90 degrees of flexion and is passively internally rotated to end-range with overpressure, reproducing the patient's pain.
* 2c. Pain with active shoulder elevation in the scapular plane.
* 2e. Pain with resisted isometric abduction.
* 2f. A history of pain in the superior part of lateral arm.
* 3. Demonstration of a painful arc of the arm from 60 to 120 of flexion

Exclusion Criteria:

* 1. Diagnosis of internal shoulder impingement.
* 2. A history of traumatic onset of shoulder pain.
* 3. Recent trauma of shoulder.
* 4. Torn tendons.
* 5. Ligamentous laxity based on a positive Sulcus and apprehension tests.
* 6. Numbness or tingling in the upper extremity
* 7. Cervical discogenic problems.
* 8. Previous shoulder or cervical spine surgery.
* 9. Systemic illness.
* 10. Corticosteroid injection on the shoulder within 1 year of the study.
* 11. Evidence of central nervous system involvement, or the inability to comply with treatment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Shoulder pain severity using the Arabic version of Shoulder Pain and Disability Index (SPADI) | baseline
  Pain domain of SPADI (pain symptoms, 5 items): each item will be scored on a visual analogue scale ranging from 0 to 10, where 0 no pain and 10 worst pain imaginable. Total pain score: ….. / 50 x 100 = % Total percentage score ranging from 0 to 100, where 0 best and 100 worst.
Shoulder disability using the Arabic version of Shoulder Pain and Disability Index (SPADI) | baseline
  Disability domain of SPADI (physical function, 8 items): each item will be scored on a visual analogue scale ranging from 0 to 10, where 0 no difficulty and 10 so difficult require help. Total disability score: ….. / 80 x 100 = % Total percentage score ranging from 0 to 100, where 0 best and 100 worst.
Measuring of scapular upward rotation angle using two bubble inclinometer | baseline
  Scapular upward rotation will be measured by using two bubble inclinometers. All patients will be assessed in a relaxed, standing (barefoot) position. One inclinometer is Velcro taped perpendicular to the humeral shaft, just above the humeral epicondyle. The resting position of the humerus will be recorded. The other inclinometer will be placed on the superior border of the spine of the scapula. Next, the patient will instruct to perform shoulder abduction to 100° with full elbow extension, neutral wrist flexion/extension and with the thumb leading to ensure vertical alignment of the inclinometer.
  When the inclinometer placed on the humerus reached 100°, the therapist records the degree of scapular upward rotation from the inclinometer placed on the spine of the scapula, each patient will perform one test, and then the measurement will recorded.
Measuring isometric scapular muscle strength using handheld dynamometer (HHD) then calculation of Upper Trapezius/Serratus Anterior strength ratio | baseline
  Upper trapezius isometric strength testing:
  The patient will seat, and the dynamometer will be placed over the superior scapula. The patient then will be asked to elevate the shoulder against resistance.
  Serratus anterior isometric strength testing:
  The patient will lay supine with the elbow and shoulder in 90° flexion. The resistance will be applied to the ulna at the olecranon process along the humeral axis. For measurement of the ratio, the isometric strength of both upper trapezius and serratus anterior will be assessed using hand-held dynamometer (HHD) and then the UT/SA ratio will be calculated. Strength = ((HHD reading in Newtons) x (distance)) Bodyweight in kilograms